CLINICAL TRIAL: NCT03772756
Title: Endoscopic Ultrasound Guided Radiofrequency Ablation (EUS-RFA) for Unresectable Pancreatic Adenocarcinoma - a Randomised Controlled Trial
Brief Title: EUS-RFA for Unresectable Pancreatic Ductal Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Jianfeng Yang, Associate director of gastroenterology department, First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-139-01
Record Dates: First submitted 2018-12-09; First posted 2018-12-11 (Actual); Last update posted 2021-08-30 (Actual); Status verified 2021-08

CONDITIONS: Pancreatic Adenocarcinoma Non-resectable
Keywords: pancreatic adenocarcinoma; radiofrequency ablation; Endoscopic ultrasound
MeSH Terms: interventions — Chemoradiotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-RFA group (Experimental): Patients in EUS-RFA group will undergo endoscopic ultrasound guided radiofrequency ablation(EUS-RFA ) and chemoradiotherapy
  Interventions: Procedure: Endoscopic ultrasound guided radiofrequency ablation; Radiation: chemoradiotherapy
- control group (Active Comparator): the control group will receive chemoradiotherapy only
  Interventions: Radiation: chemoradiotherapy

INTERVENTIONS:
Procedure: Endoscopic ultrasound guided radiofrequency ablation — Endoscopic ultrasound guided radiofrequency ablation （EUS-RFA） will be done in 3 different sessions with 2 weeks interval between each session on Day 1, Day 15 and Day 30. Each session will involve multiple applications of EUS-RFA (up to 10) with RF setting of 25 Watts over 90 seconds for each application.
  Other Names: EUS-RFA
  Arms: EUS-RFA group
Radiation: chemoradiotherapy — Receive chemoradiotherapy

SUMMARY:
the study evaluate the efficacy and safety of EUS-RFA using Habib EUS-RFA catheter with a prospective randomised trial in patients with inoperable PDAC.

DETAILED DESCRIPTION:
The five year survival for pancreatic ductal adenocarcinoma (PDAC) is less than 5% in spite of the advances in management of cancers in the last few decades. Endobiliary application of radiofrequency ablation (RFA) has been developed in our unit and used in patients with unresectable bile duct and pancreatic head adenocarcinomas presenting with biliary obstruction. Various techniques of EUS-guided tumour ablation have been described, including RF ablation, photodynamic therapy, laser ablation, and ethanol injection. Endoscopic ultrasound guided RFA (EUS-RFA) of the pancreatic head using Habib EUS-RFA catheter through a 19-gauge needle was well tolerated in 5 Yucatan pigs and with minimum amount of pancreatitis .

ELIGIBILITY:
Inclusion Criteria:

* Patients in the age group 20 to 80 years
* A cytological or histological diagnosis of inoperable PDAC based on multidisciplinary review of cross sectional imaging and cytology or histology results.
* Patients who have been deemed unfit for surgical resection of the PDAC subjects who are fit for surgical resection but have declined surgery will also be considered for the study
* PDAC patients presenting with jaundice to be considered after a successful biliary drainage
* Patients ought to be fit enough to be considered for the study (ECOG performance status 0, 1 or 2)
* Patients capable of giving informed consent

Exclusion Criteria:

* Inability to give informed consent
* Pregnancy or breast feeding
* ECOG performance status 3 or 4
* Life expectancy less than 3 months
* Patients with distant metastases or malignant ascites

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-12-20 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-16 (Actual)

PRIMARY OUTCOMES:
Change in tumour size as measured on EUS and or CT | 60 days
  The tumor size was compared before and after 60 days EUS-RFA
Change in serum levels of Ca 19-9 | 60 days
  Serum levels of Ca 19-9 was compared before and after 60 days EUS-RFA

SECONDARY OUTCOMES:
Overall survival at 6 months | 6 months
  Survival rate 6 months after EUS-RFA
Overall survival at 12 months | 12 months
  Survival rate 12 months after EUS-RFA

CONTACTS AND LOCATIONS:
Overall Officials: Xiaofeng Zhang, Principal Investigator — First People's Hospital of Hangzhou
Locations (2):
- China (2):
  - Jianfeng Yang, Hangzhou, Zhejiang
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang

REFERENCES:
- [Background] Gaidhane M, Smith I, Ellen K, Gatesman J, Habib N, Foley P, Moskaluk C, Kahaleh M. Endoscopic Ultrasound-Guided Radiofrequency Ablation (EUS-RFA) of the Pancreas in a Porcine Model. Gastroenterol Res Pract. 2012;2012:431451. doi: 10.1155/2012/431451. Epub 2012 Sep 20. PMID 23049547